CLINICAL TRIAL: NCT05651126
Title: Modulation of Serotonin Pathways Using Psilocybin in Adults With and Without Autism Spectrum Disorder (ASD)
Brief Title: Psilocybin in Adults With and Without Autism Spectrum Disorder
Acronym: PSILAUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Grainne McAlonan, Deputy Head of Department, King's College London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRAS: 292281; REC: 21/LO/0795
Record Dates: First submitted 2022-11-11; First posted 2022-12-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Psilocybin; Serotonin; Pharmacological Imaging; MRI; EEG; Psychedelics
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Case-Control comparison using repeated-measures cross-over design. Each participant receives each one of the three pharmacological probes in separate visits (i.e., placebo, psilocybin low dose and psilocybin higher dose), with the order of administration being pseudorandomized (to prevent order effects).
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded to the drug condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo, Psilocybin_2, Psilocybin_5 (Experimental): Dose order: Placebo, Psilocybin 2mg, Psilocybin 5mg
  Interventions: Drug: Psilocybin 5 mg; Drug: Psilocybin 2 mg; Drug: Placebo
- Psilocybin_2, Placebo, Psilocybin_5 (Experimental): Dose order: Psilocybin 2mg, Placebo, Psilocybin 5mg
  Interventions: Drug: Psilocybin 5 mg; Drug: Psilocybin 2 mg; Drug: Placebo
- Psilocybin_2, Psilocybin_5, Placebo (Experimental): Dose order: Psilocybin 2mg, Psilocybin 5mg, Placebo
  Interventions: Drug: Psilocybin 5 mg; Drug: Psilocybin 2 mg; Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin 5 mg — Partial Serotonin (5HT) 1A/2A Receptor Agonist Psilocybin
  Other Names: COMP360
Drug: Psilocybin 2 mg — Partial Serotonin (5HT) 1A/2A Receptor Agonist Psilocybin
  Other Names: COMP360
Drug: Placebo — Inactive placebo

SUMMARY:
This study will test the hypothesis that brain systems are differentially regulated by serotonin in individuals with and without Autism Spectrum Disorder.

DETAILED DESCRIPTION:
To do this, the brain response to two single acute doses of partial serotonin (5HT)1A/2A receptor agonist psilocybin (COMP360) relative to a single dose of placebo (baseline serotonin activity) will be compared in healthy autistic and non-autistic adults.

Brain function will be assessed using a range of MRI (fMRI and MRS), EEG and sensory tasks. Unimodal and multimodal analyses will be conducted.

Please note that this study uses psilocybin as a probe of the serotonin system in a Case-Control science study and, following Scope protocol review, the U.K. MHRA confirmed that it is not a 'Clinical Trial of an Investigational Medicinal Product' (IMP) as defined by the EU Directive 2001/20/EC.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Calendar age above 18 years
* Working knowledge of English
* Able to give informed consent
* Not pregnant or breastfeeding
* Individuals should be in good physical health, prescription medication free during the 2-week period preceding a study visit. However, occasional use of over-the-counter medication (e.g. painkillers) on an as needed basis (and not on the day of study visit) may be permitted. In addition, regular prescription medication (use of a stable dose over the two months preceding participation) with a drug that does not affect 5HT directly may be permitted. Also permitted is topical medication without systemic exposure

For individuals with ASD:

* Diagnosis of ASD by recognised clinical service supported by the Autism Diagnostic Interview-Revised (ADI-R) if a relative is available. Current symptom level assessed using the Autism Diagnostic Observation Schedule (ADOS-2)

Exclusion Criteria:

For all participants:

* History of allergy/idiosyncrasy to psilocybin or chemically related compounds or excipients which may be employed in the study or to any other drug used in the past
* Clinically relevant history or presence of any medical disorder, potentially interfering with this study
* Clinically relevant abnormality at screening as judged by the investigator
* History of or current abuse of drugs (including prescription medication) or alcohol or solvents
* Participation in a research study involving a pharmacological probe or drug trial within last month
* Subjects with current epilepsy, seizures or episodes of unexplained and unprovoked loss of consciousness
* Anyone with a history or examination which indicates laboratory testing is needed will be excluded from the study
* Intelligence Quotient below 70
* Currently taking prescription medications of propranolol or pindolol
* Individuals with major mental illness
* Individuals who have a current or past history of meeting diagnostic criteria for schizophrenia or other psychotic disorders or bipolar I or II disorder

Reproductive safety:

* Pregnancy or breastfeeding (is a routine exclusion for research MRI scanning)
* Female study participants must be willing to use one form of highly effective non-hormonal contraception for one week after study drug administration. This would include a vasectomised partner (sole partner), tubal occlusion, intrauterine system [IUS]/hormonal coil or copper containing intrauterine device or copper containing IUD, or true abstinence (when this is in line with the preferred and usual lifestyle of the subject). Women should have been stable on their chosen method of birth control for a minimum of 2 months before entering the study. Participants must agree to undergo a pregnancy test prior to each administration of study drug

For individuals with ASD:

ASD caused by a known genetic syndrome, e.g. Fragile X, 22q11 deletion syndrome.

Currently treated for epilepsy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Brain activation and connectivity response to serotonergic stimulation as assessed by functional magnetic resonance imaging. | Data collected on up to 3 visit days per participant.
  Comparing whole brain blood-oxygen-level-dependent (BOLD) activation (institutional units) during the resting state in cases and controls when the serotonin system is activated by a single oral dose of psilocybin (COMP360) versus the placebo condition.
Brain electrophysiological activity task-free electroencephalography (EEG) | Data collected on up to 3 visit days per participant.
  Case-control comparison of task-free EEG by time-frequency analysis during placebo and when serotonin system is activated with psilocybin.
Brain electrophysiological activity electroencephalography (EEG) during visual stimulation | Data collected on up to 3 visit days per participant.
  Case-control comparison of EEG Evoked Potentials in response to visual stimulation during placebo and when serotonin system is activated with psilocybin.
Brain electrophysiological activity electroencephalography (EEG) during auditory stimulation | Data collected on up to 3 visit days per participant.
  Case-control comparison of EEG Event Related Potentials in response to auditory tones during placebo and when serotonin system is activated with psilocybin.

SECONDARY OUTCOMES:
Brain excitation and inhibition response to serotonergic stimulation as assessed by magnetic resonance spectroscopy. | Data collected on up to 3 visit days per participant.
  Quantification and case-control comparison of brain metabolites relevant to regulation of excitation and inhibition (focus on Glx, GABA, GSH) using proton magnetic resonance spectroscopy when serotonin system is 'at rest' (placebo) and when activated by psilocybin.

OTHER OUTCOMES:
Exploratory: Subjective effects intensity | Data collected on up to 3 visit days per participant.
  5-Dimensional altered states of consciousness (5D-ASC) used for Case-control comparison of subjective effects intensity at placebo and when serotonin system activated with psilocybin

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whelan TP, Daly E, Puts NA, Smith P, Allison C, Baron-Cohen S, Malievskaia E, Murphy DGM, McAlonan GM. The 'PSILAUT' protocol: an experimental medicine study of autistic differences in the function of brain serotonin targets of psilocybin. BMC Psychiatry. 2024 Apr 25;24(1):319. doi: 10.1186/s12888-024-05768-2. PMID 38658877